CLINICAL TRIAL: NCT04739683
Title: Cervical Ripening With Foley Bulb Versus Dilapan-S at Home: a Randomized Trial
Brief Title: Cervical Ripening With Foley Bulb Versus Dilapan-S at Home
Acronym: GOHOME
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to another study which superseded it.
Sponsor: Christiana Care Health Services (Other)
Collaborators: Medicem International CR s.r.o. (Industry); Medicem Technology s.r.o. (Other)
Responsible Party: Principal Investigator, Anthony Sciscione, DO, Physician-Perinatology, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDD#604684
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Induced; Birth; Induction of Labor Affected Fetus / Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Foley bulb (Active Comparator): 16F latex or silicone Foley catheter inflated with 30-40 cc of sterile water. The catheter will be taped to the inner thigh with gentle traction.
  Interventions: Device: Foley bulb placement
- DILAPAN-S® (Active Comparator): Synthetic hydrogel cervical dilator consists of the dilating part, the polypropylene handle, and the marker string. The dilating part is manufactured from an anisotropic xerogel of AQUACRYL.
  Interventions: Device: DILAPAN-S® placement

INTERVENTIONS:
Device: Foley bulb placement — A 16 F Foley catheter with a 30-mL balloon and stylet is inserted into the endocervical canal under direct visualization by sterile speculum exam or by digital palpation. The Foley catheter is advanced to or past the internal os, and the balloon is filled with 30-40 mL of sterile water. The catheter is then placed on genital traction by taping the end of the catheter to the medial portion of the thigh.
  Arms: Foley bulb
Device: DILAPAN-S® placement — A bivalve speculum will be used to visualize and prepare the cervix with an antiseptic solution. The DILAPAN-S® (4 x 65 mm) will be inserted in the cervical canal until it traverses the internal os. As many dilators as needed to achieve the desired effect should be inserted. Specific number of pieces always depends on decision and clinical judgement of physician and indications. A gauze pad moistened with sterile water or saline may be inserted into the vagina to help keep the DILAPAN-S® in place, if needed
  Arms: DILAPAN-S®

SUMMARY:
DILAPAN-S® was FDA-approved for pre-induction cervical ripening in 2015. Since that time, there have been limited studies comparing its efficacy, safety, and patient satisfaction to other mechanical cervical ripening techniques. The purpose of this trial is to perform a noninferiority randomized clinical trial comparing DILAPAN-S® to the Foley catheter for outpatient cervical ripening in term elective labor inductions, examining time spent on the labor and delivery unit, patient safety, and patient satisfaction feedback.

DETAILED DESCRIPTION:
In 2019, Grobman et al, published the ARRIVE trial showing that labor inductions without medical indication at 39 weeks gestation are associated with improved maternal and perinatal outcomes compared to expectant management.1 In the wake of these landmark findings, labor inductions without medical indication are becoming increasingly common not only on a nation scale, but locally as well. Recent data show that labor inductions without medical indication encompass nearly one third of all inductions at Christiana Care Health System.

Labor induction can include both mechanical and pharmacological measures to ripen the cervix and stimulate uterine contractions. The ultimate challenge, which has been the focus of numerous studies to date, is to determine which mechanical and/or pharmacological products and which clinical settings are safest and most efficacious for inducing labor.

Currently, transcervical Foley catheters are the gold-standard mechanical method of cervical ripening. However, new-emerging data has shown that hygroscopic cervical dilators, traditionally used for early pregnancy termination, may be a viable alternative. DILAPAN-S® , a hygroscopic dilator composed of a synthetic hydrogel was approved by the Food and Drug Administration for cervical ripening in 2015 and has been the subject of recent investigation. In a single-center, randomized, open-label trial consisting of 419 patients, Saad et al showed that DILAPAN-S® is not inferior to the Foley catheter for pre-induction cervical ripening at term; there was no significant difference in maternal and neonatal adverse events and patients with DILAPAN-S® were more satisfied than patients with the Foley catheter as far as sleep, relaxing time, and performance of desired daily activities.2

Furthermore, in the pursuit of improving patient satisfaction with consideration of healthcare resources, studies have investigated the safety and efficacy of outpatient mechanical cervical ripening.3 Sciscione et al, showed that in a low-risk population of 1,905 patients, no adverse outcomes were associated with outpatient Foley catheter cervical ripening and patients on average avoided 9.6 hours of hospitalizations compared to the inpatient group.4 The ACOG practice bulletin on induction of labor now states that outpatient cervical ripening, particularly mechanical methods, may be appropriate in select patients.5 Based on the literature cited above, it is plausible to hypothesize that DILAPAN-S® used for outpatient cervical ripening may optimize patient satisfaction and healthcare resource utilization without compromising patient safety and efficacy. The purpose of this trial is to perform a noninferiority randomized clinical trial comparing DILAPAN-S® to the Foley catheter for outpatient cervical ripening in term elective labor inductions, examining time spent on the labor and delivery unit, patient safety, and patient satisfaction feedback.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation. Twin gestation reduced to singleton, either spontaneously or therapeutically is not eligible unless the reduction occurred before 14 weeks 0 days gestational age.
* Gestational age at randomization between 39 weeks and 40 weeks 6 days (based on reliable EGA defined as ultrasound performed before 14 weeks 0 days, or a certain LMP consistent with ultrasonography before 21 weeks and 0 days.)
* Patient prefers outpatient cervical ripening
* Patient lives within a one-hour commute from the hospital.

Exclusion Criteria:

* Project gestational age at date of first ultrasound is > 20 weeks 6 days
* Refusal of blood products
* Participation in another interventional study that influences management of labor at delivery or perinatal morbidity or mortality
* Delivery planned elsewhere at a non-Christiana site
* Major maternal medical illness associated with increased risk for adverse pregnancy outcomes that would preclude her from an outpatient induction (e.g. any diabetes mellitus, lupus, any hypertensive disorder, cardiac disease, renal insufficiency)
* Medical indication for induction prior to 40 weeks 5 days due to any maternal
* Heparin or low-molecular weight heparin use during the current pregnancy
* Cerclage in current pregnancy
* Prior uterine or cervical surgery (cesarean, myomectomy, cerclage, LEEP, cone biopsy, etc.)
* Known HIV positivity because of modified delivery plan
* Iodine or latex allergy
* Fetal demise or known major fetal anomaly
* Medical indication for induction prior to 40 weeks 5 days due to any fetal condition
* Known oligohydramnios, defined as amniotic fluid index < 5 cm or maximal vertical pocket < 2 cm
* Fetal growth restriction, defined as EFW < 10th percentile
* Plan for cesarean delivery or contraindication to labor
* Nonvertex fetal presentation
* Placenta previa, placenta accrete, or vasa previa
* Active genital herpes lesions
* Cervical dilation greater than 3 cm on initial evaluation
* Signs of labor (regular painful contractions with cervical change) on initial evaluation
* Active vaginal bleeding greater than bloody show on initial evaluation
* Ruptured membranes on initial evaluation
* Non-reassuring fetal status (category II or III fetal heart rate tracing) on initial evaluation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Time spent on the labor and delivery unit | through study completion, an average of 2 years
  Length of time spent on the labor and delivery unit, hours

SECONDARY OUTCOMES:
Rate of vaginal delivery | through study completion, an average of 2 years
Rate of cesarean delivery | through study completion, an average of 2 years
Indication for cesarean delivery | through study completion, an average of 2 years
  Reasons for cesarean delivery include: non-reassuring fetal heart rate tracing, arrest of dilation, arrest of descent, failed induction of labor, maternal request, other
Time from device insertion to delivery | through study completion, an average of 2 years
  Time from device (Foley bulb or Dilapan) insertion to delivery (vaginal or cesarean), hours
Rate of vaginal delivery within 24 hours of device insertion | through study completion, an average of 2 years
Rate of vaginal delivery within 36 hours of device insertion | through study completion, an average of 2 years
Time from device insertion to expulsion or extraction | through study completion, an average of 2 years
  Time from device (Foley bulb or Dilapan) insertion to spontaneous expulsion or device removal, hours
Rate of device expulsion at home | through study completion, an average of 2 years
  Percentage of patients whose device (Foley bulb or Dilapan) was expelled at home
Rate of patients that received Pitocin | through study completion, an average of 2 years
Average number of Dilapan dilator rods used | through study completion, an average of 2 years
  Multiple Dilapan rods may be placed for cervical dilation. The number of rods used is at the discretion of the clinician.
Change in Bishop score before and after mechanical cervical ripening | through study completion, an average of 2 years
  Change in Bishop score from initial assessment to first exam following device expulsion/removal.
Time from device insertion to active stage of labor | through study completion, an average of 2 years
  The active stage of labor is defined as cervical dilation greater than or equal to 6cm, hours
Rate of artificial rupture of membranes | through study completion, an average of 2 years
Rate of epidural or spinal anesthesia during labor | through study completion, an average of 2 years
Rate of analgesia needed for device insertion | through study completion, an average of 2 years
  Analgesia methods may include butorphanol, neuraxial blockade, nitric oxide, etc.
Rate of complications from device insertion | through study completion, an average of 2 years
  Complications include: incidental rupture of membranes, device malfunction/breakage, vaginal bleeding (defined as gross blood apparent on glove, perineum, vagina, or within Foley catheter lumen), cervical laceration, vasovagal reaction
Rate of tachysystole | through study completion, an average of 2 years
  Defined as at least 6 contractions in 10 minutes for 2 consecutive 10-minute periods
Rate of postpartum hemorrhage | through study completion, an average of 2 years
  Defined as 1,000 mL or blood loss accompanied by signs or symptoms of hypovolemia within 24 hours after the birth process
Rate of shoulder dystocia | through study completion, an average of 2 years
Rate of suspected intraamniotic infection | through study completion, an average of 2 years
  Defined as the presence of maternal intrapartum fever and one or more of the following: maternal leukocytosis, purulent cervical drainage, or fetal tachycardia
Rate of any serious maternal morbidity | through study completion, an average of 2 years
  Serious maternal morbidities include uterine rupture, admission to an intensive care unit, and sepsis
Rate of maternal death | through study completion, an average of 2 years
Maternal satisfaction | through study completion, an average of 2 years
  A two-part maternal satisfaction survey will be administered immediately after device placement and then postpartum day one
Rate of 1 minute Apgar score < 5 | through study completion, an average of 2 years
  Rate of 1 minute Apgar score less than 5
Rate of 5 minute Apgar score < 7 | through study completion, an average of 2 years
  Rate of 5 minute Apgar score less than 7
Rate of NICU admission | through study completion, an average of 2 years
  Rate of neonates admitted to the NICU
Rate of NICU admission > 48 hours | through study completion, an average of 2 years
  Rate of neonates requiring NICU admission for longer than 48 hours
NICU length of stay | through study completion, an average of 2 years
  Length of NICU admission, days
Rate of any adverse neonatal outcome | through study completion, an average of 2 years
  Includes death, severe respiratory distress syndrome (defined as intubation and mechanical ventilation for a minimum of 12 hours), hypoxic-ischemic encephalopathy, seizure, culture-proven neonatal sepsis, birth trauma (bone fracture, intracranial hemorrhage, neurologic injury, retinal hemorrhage), hypotension requiring vasopressor support, receipt of total body cooling.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony C Sciscione, DO, Principal Investigator — Christiana Care Health Services

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Saad AF, Villarreal J, Eid J, Spencer N, Ellis V, Hankins GD, Saade GR. A randomized controlled trial of Dilapan-S vs Foley balloon for preinduction cervical ripening (DILAFOL trial). Am J Obstet Gynecol. 2019 Mar;220(3):275.e1-275.e9. doi: 10.1016/j.ajog.2019.01.008. Epub 2019 Feb 18. PMID 30790569
- [Background] Levine LD, Sciscione AC. Foley Catheter for Outpatient Cervical Ripening: Review of the Evidence and a Proposed Model of Care. Am J Perinatol. 2019 Dec;36(14):1528-1532. doi: 10.1055/s-0038-1677473. Epub 2019 Jan 23. No abstract available. PMID 30674049
- [Background] Sciscione AC, Bedder CL, Hoffman MK, Ruhstaller K, Shlossman PA. The timing of adverse events with Foley catheter preinduction cervical ripening; implications for outpatient use. Am J Perinatol. 2014 Oct;31(9):781-6. doi: 10.1055/s-0033-1359718. Epub 2013 Dec 17. PMID 24347259
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Albers LL. The duration of labor in healthy women. J Perinatol. 1999 Mar;19(2):114-9. doi: 10.1038/sj.jp.7200100. PMID 10642971